CLINICAL TRIAL: NCT05544032
Title: Expanded Access of Axatilimab to Treat a Single Patient With Chronic Graft Versus Host Disease (GVHD)
Status: Available | Type: Expanded Access
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: I-34176-25-07
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Chronic Graft Vs. Host Disease
Keywords: Chronic Graft Vs. Host Disease; cGVHD
MeSH Terms: interventions — axatilimab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: axatilimab — Treatment with axatilimab includes receiving intravenous (IV) doses of axatilimab every 2 weeks
  Other Names: INCA34176

SUMMARY:
This program is being offered on a patient by patient basis and will require company, Institutional Review Board/Independent Ethics Committee and Single Patient IND approval.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult